CLINICAL TRIAL: NCT05485337
Title: Effectiveness of Therapeutic Tactics of Analgesia in Patients With Gunshot and Mine-explosive Wounds at the Stages of Treatment
Acronym: ETTAPGM-EWST
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Vasyl' Horoshko, Chief researcher, Bogomolets National Medical University
Other Study IDs: №158/23/05/2022
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Chronic Pain
Keywords: pain treatment, analgesia, wounds, stages of treatment.
MeSH Terms: conditions — Chronic Pain; Agnosia; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective analysis: A retrospective analysis of disease histories for the period from 2014 to 2021 was carried out. Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
  Interventions: Other: visual analog scale
- prospective study: Recruitment of patients for the prospective study was carried out in the period from 02.24.2022 to 05.24.2022
  Interventions: Other: visual analog scale

INTERVENTIONS:
Other: visual analog scale — Data collection was carried out at all stages of treatment: medical and nursing brigade, military mobile hospital, military medical clinical center, during rehabilitation, within 12 months of the injury.
  Other Names: neuropathic pain Didier Bouhassiraa, Nadine Attala et al. Pain, 2005, 114: 29-36 (DN4).; Chaban Quality of Life Scale; The Hospital Anxiety and Depression Scale (HADS); Mississippi PTSD scale (military version)

SUMMARY:
In 82.1% of patients with gunshot and mine-explosive wounds, pain becomes chronic, therefore, the study of the effectiveness of therapeutic tactics for pain relief in this category of patients at the stages of treatment will be important for improving the results of pain treatment.

DETAILED DESCRIPTION:
The effectiveness of the therapeutic tactics of analgesia in patients with gunshot and mine-explosive wounds at the stages of treatment needs to be studied, because the subjective feelings and emotional experiences experienced by patients during the wounding in combat conditions through the prism of psychological disorders have their own characteristics. Given that in 82.1% of cases it is not possible to achieve a positive result of treatment, the data of our study will play an important role in their treatment.

ELIGIBILITY:
Inclusion Criteria:

* the presence of gunshot wounds

Exclusion Criteria:

* no gunshot wounds

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients were injured during hostilities
Sampling Method: Probability Sample
Enrollment: 2215 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 12 months
  from 0 to 10 points
Didier Bouhassiraa DN4 | 12 months
  4 or more points (a neuropathic pain component is present)
The Hospital Anxiety and Depression Scale | 12 months
  0-7 is the norm 8-13 - mild depressive disorders 14-18 - depressive disorders of medium severity 19-22 - severe depressive disorders 23 and more - depressive disorders of a very severe degree of severity
Chaban Quality of Life Scale | 12 months
  up to 56 inclusive - a very low level 57-66 - low 67-75 - average 76-82 - tall 83-100 is very high
Mississippi PTSD scale (military version) | 12 months
  the mean values of the total score are 76±18 for well-adjusted servicemen, 86±26 for servicemen with mental disorders, and 130±18 for those with PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Bogomolets National Medical University, Ministry of Health of Ukraine, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided
I plan to share